CLINICAL TRIAL: NCT01966289
Title: A Pilot Study of SGI-110 in Combination With an Allogeneic Colon Cancer Cell Vaccine (GVAX) and Cyclophosphamide (CY) in Metastatic Colorectal Cancer (mCRC) as Maintenance Therapy
Brief Title: SGI-110 in Combination With an Allogeneic Colon Cancer Cell Vaccine (GVAX) and Cyclophosphamide (CY) in Metastatic Colorectal Cancer (mCRC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Astex Therapeutics, Ltd (Unknown); Susan Cohan Colon Cancer Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J13138; NA_00087578 (Other: JHMIRB)
Record Dates: First submitted 2013-10-10; First posted 2013-10-21 (Estimated); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Colorectal Neoplasms; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Neoplasms; Digestive System Diseases; Gastrointestinal Diseases; Colonic Diseases; Intestinal Diseases; Rectal Diseases
MeSH Terms: conditions — Colorectal Neoplasms; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Neoplasms; Digestive System Diseases; Gastrointestinal Diseases; Colonic Diseases; Intestinal Diseases; Rectal Diseases | interventions — Cyclophosphamide; guadecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 1:CY/GVAX concurrently with SGI-110 (Experimental): During each of the four cycles, Cyclophosphamide (CY) is administered on Day 1 at 200 mg/m2, the colon cancer tumor vaccine (GVAX) is administered on Day 2 at 5E8 colon cancer cells + 5E7 Granulocyte macrophage-colony stimulating factor (GM-CSF) secreting cells, and SGI-110 is administered on Days 1-5 at 60 mg/m2. Each cycle is 28 days. Enrollment will begin first in Cohort 1 and 2. If a response to the treatment is seen in Cohorts 1 and 2, enrollment in Cohort 3 and 4 will begin.
  Interventions: Drug: CY; Biological: GVAX; Drug: SGI-110
- Cohort 2: CY/GVAX after SGI-110 (Experimental): During each of the four cycles, SGI-110 is administered on Days 1-5 at 60 mg/m2, Cyclophosphamide (CY) is administered on Day 8 at 200 mg/m2, and the colon cancer tumor vaccine (GVAX) is administered on Day 9 at 5E8 colon cancer cells + 5E7 GM-CSF secreting cells. Each cycle is 28 days. Enrollment will begin first in Cohort 1 and 2. If a response to the treatment is seen in Cohorts 1 and 2, enrollment in Cohort 3 and 4 will begin.
  Interventions: Drug: CY; Biological: GVAX; Drug: SGI-110
- Cohort 3: CY/GVAX (Experimental): During each of the four cycles, Cyclophosphamide (CY) is administered on Day 1 at 200 mg/m2 and the colon cancer tumor vaccine (GVAX) is administered on Day 2 at 5E8 colon cancer cells + 5E7 GM-CSF secreting cells. Each cycle is 28 days. Enrollment will begin first in Cohort 1 and 2. If a response to the treatment is seen in Cohorts 1 and 2, enrollment in Cohort 3 and 4 will begin.
  Interventions: Drug: CY; Biological: GVAX
- Cohort 4: SGI-110 (Experimental): During each of the four cycles, SGI-110 is administered on Days 1-5 at 60 mg/m2. Each cycle is 28 days. Enrollment will begin first in Cohort 1 and 2. If a response to the treatment is seen in Cohorts 1 and 2, enrollment in Cohort 3 and 4 will begin.
  Interventions: Drug: SGI-110

INTERVENTIONS:
Drug: CY — CY is administered intravenously at 200 mg/m2
  Other Names: Cyclophosphamide, Cytoxan
  Arms: Cohort 1:CY/GVAX concurrently with SGI-110; Cohort 2: CY/GVAX after SGI-110; Cohort 3: CY/GVAX
Biological: GVAX — GVAX is administered intradermally at 5E8 colon cancer cells + 5E7 GM-CSF secreting cells
  Other Names: Colon cancer tumor vaccine
  Arms: Cohort 1:CY/GVAX concurrently with SGI-110; Cohort 2: CY/GVAX after SGI-110; Cohort 3: CY/GVAX
Drug: SGI-110 — SGI-110 is administered subcutaneously at 60 mg/m2
  Arms: Cohort 1:CY/GVAX concurrently with SGI-110; Cohort 2: CY/GVAX after SGI-110; Cohort 4: SGI-110

SUMMARY:
This study will be looking at whether CY/GVAX in combination with SGI-110 is effective (recruits CD45RO+ T cells to the tumor which may be a marker of anti-tumor activity) and safe in patients with metastatic colon or rectum cancers.

ELIGIBILITY:
Inclusion Criteria:

1. Documented cancer of the colon or rectum who have received and are stable on first or second-line therapy regimens for metastatic colorectal cancer
2. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 1
3. Adequate organ function as defined by study-specified laboratory tests
4. Must use acceptable form of birth control through the study and for 28 days after final dose of study drug
5. Signed informed consent form
6. Willing and able to comply with study procedures

Exclusion Criteria:

1. Currently have or have history of certain study-specified heart, liver, kidney, lung, neurological, immune or other medical conditions
2. Systemically active steroid use
3. Another investigational product within 28 days prior to receiving study drug
4. Major surgery or significant traumatic injury (or unhealed surgical wounds) occurring within 28 days prior to receiving study drug
5. Chemotherapy, radiation, hormonal, or biological cancer therapy within 28 days prior to receiving study drug
6. Pregnant or lactating
7. Unwilling or unable to comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-04-14 (Actual); Primary Completion 2020-06-06 (Actual); Study Completion 2020-06-06 (Actual)

PRIMARY OUTCOMES:
Difference in CD45RO+ tumor infiltrating lymphocytes (TILs) measured by immunohistochemistry in pre and post-treatment tumor biopsies from patients with metastatic colorectal cancer | 4 years
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 4 years

SECONDARY OUTCOMES:
Overall Survival (OS) | 4 years
Time To Progression (TTP) | 4 years
Progression Free Survival (PFS) | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Nilofer Azad, MD, Principal Investigator — The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Bever KM, Thomas DL 2nd, Zhang J, Diaz Rivera EA, Rosner GL, Zhu Q, Nauroth JM, Christmas B, Thompson ED, Anders RA, Judkins C, Liu M, Jaffee EM, Ahuja N, Zheng L, Azad NS. A feasibility study of combined epigenetic and vaccine therapy in advanced colorectal cancer with pharmacodynamic endpoint. Clin Epigenetics. 2021 Feb 2;13(1):25. doi: 10.1186/s13148-021-01014-8. PMID 33531075